CLINICAL TRIAL: NCT04017416
Title: Controlled Trial of the I-PLAN Intervention to Promote Hearing Aid Use Among First Time Adult Hearing Aid Users
Brief Title: Controlled Trial of the I-PLAN Intervention
Status: Completed | Type: Observational
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Noor Afzarini Hasnita Binti Ismail, Principle Investigator, University of Manchester
Other Study IDs: 17/NW/0406
Record Dates: First submitted 2019-07-04; First posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Hearing Aid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard Care: Audiologists in the standard care group were instructed to manage the patients in the same way as they would do in their routine clinics which were in accordance with national practice guidelines and were typical of National Healthcare Services (NHS) audiology departments across the UK.
- I-PLAN: Audiologists were instructed to deliver the I-PLAN in addition to standard care at the hearing aid fitting consultation.
  Interventions: Behavioral: I-PLAN

INTERVENTIONS:
Behavioral: I-PLAN — The I-PLAN is a behaviour change intervention that consists of; information on consequences of hearing aid use/non-use, reminder prompt and behavioural plan to promote hearing aid use.
  Groups: I-PLAN

SUMMARY:
That is a need for intervention to promote hearing aid use among adult patients with hearing aids. The aim of the present study was, for the first time, to evaluate the efficacy of the I-PLAN intervention to promote hearing aid use.

DETAILED DESCRIPTION:
The I-PLAN is a behaviour change theory-based intervention to promote hearing aid use. It consists of; 1. information on consequences of using and not using a hearing aid, 2. a physical prompt as a reminder to hearing aid use and 3. a behavioural plan to use a hearing aid. The aim of this study was to test efficacy of the I-PLAN intervention, delivered face-to-face by study audiologists. 160 first-time hearing aid users were recruited at the hearing aid fitting appointment. Adult patients were allocated either to the I-PLAN group or Standard Care group. Adult patients were allocated to the groups based on the clinic schedules of study audiologists.

ELIGIBILITY:
Inclusion Criteria:

* had no previous personal experience of using a hearing aid
* were aged 18 years old or above
* attended initial hearing aid fitting appointment with study audiologists
* were native English speakers or had good understanding of English
* had sufficient mental capacity to provide informed consent based on audiologist's opinion were eligible to take part in this study

Exclusion Criteria:

* inability to complete the questionnaires due to age-related problems (for example; dementia) based on audiologist's opinion
* presence of medical contraindications for hearing aids as described by the British Academy of Audiology (BAA 2007)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study recruited adult patients who were first-time hearing aid users.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Subjective hearing aid use based on Glasgow Hearing Aid Benefit Profile questionnaire | 6 weeks
  Self-reported hearing aid use with 5 response options (1-never/not all to 5 - all the time). Total score 5.

SECONDARY OUTCOMES:
Objective hearing aid use | 6 weeks
  Hearing aid use were measured from data-logging downloaded from hearing aid(s)
International Outcome Inventory for Hearing Aids | 6 weeks
  Self-reported hearing aid benefit with five response options (from 1 to 5). Higher score indicate better outcomes
Self-reported Hearing Handicap Inventory for the Elderly and for Adults - Screening version | 6 weeks
  Self-reported hearing aid benefit with three response options (yes- 4 points, sometimes- 2 points and no - 0 points). Higher scores indicate greater perceived hearing handicap
Self-regulation in relation to hearing aid use | 6 weeks
  Self-reported self-regulation with a seven point Likert scale (1 strongly disagree to 7 strongly agree). Higher scores indicate greater self-regulation
Habit formation | 6 weeks
  Self-reported habit formation with seven point Likert scale (1 strongly disagree to 7 strongly agree). Higher the scores indicate stronger habit

CONTACTS AND LOCATIONS:
Overall Officials: Piers Dawes, PhD, Principal Investigator — Manchester Centre for Audiology and Deafness
Locations (1):
- Audiology Clinic, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided